CLINICAL TRIAL: NCT00211731
Title: Improving the Delivery of Effective Care to Minorities
Brief Title: Preventing Recurrent Stroke in Minority Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-0053; P01HS010859-05 (AHRQ)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2007-12

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: Acute stroke; recurrent stroke preventive measures; racial disparities
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

INTERVENTIONS:
Behavioral: Chronic Disease Self Management Course

SUMMARY:
This study focuses on causes of under-use of secondary stroke preventive measures demonstrated in randomized clinical trials to be efficacious, but not appropriately utilized in urban, minority populations.

DETAILED DESCRIPTION:
As the population ages and the number of prevalent strokes increases recurrent stroke is becoming an increasingly important health care burden. National and local data strongly suggest that this burden falls disproportionately on minority populations, notably Blacks and Hispanics. This study seeks to determine the factors that contribute to that disparity and design and implement a novel intervention tailored to alleviate the factors identified. Specifically it will focus on causes of under-use of stroke preventive measures demonstrated in randomized clinical trials to be efficacious, but not appropriately utilized in urban, minority populations.

In the first phase of the study, charts of acute stroke patients in 4 large urban hospitals that serve the 3 racial/ethnic groups under study (Blacks, Hispanics and non-Hispanic whites) will be reviewed to determine the magnitude of under-use of these measures. Simultaneously, a panel of local expert physicians will finalize the proposed criteria for appropriate attention to risk factor assessment and modification. In the second phase of the proposed work, we will conduct a randomized trial intervention strategy that will include a control arm, and a patient educational arm where participants will be enrolled in a Chronic Disease Self Management Program. The program is designed to teach patients tools for managing their chronic illness which will empower them to improve their overall health. The program will be specifically tailored for patients living with asymptomatic chronic illnesses and will emphasize communication with health care providers. The educational intervention will be accompanied by a two-phased chart abstraction to measure clinical markers pre and post intervention. In the final phase of the study, the results of the trial will be analyzed and the results disseminated

ELIGIBILITY:
Inclusion Criteria:

Non-Hispanic white, Non-Hispanic Black or Hispanic patients hospitalized at one of the four participating hospitals for acute stroke or TIA or rehabilitation immediately following an acute stroke. Patients must speak English or Spanish, must be able to communicate verbally, and must be cognitively aware and able to participate in group discussions.

Exclusion Criteria:

This study is about racial and ethnic disparities regarding recurrent stroke in Non-Hispanic white, Non-Hispanic Black and Hispanic populations. The study does not include other races. We are excluding anyone who is under 40 years old because the etiology of stroke for these patients is different than older patients. Patients will be excluded who had a stroke secondary to substance abuse or who had an intra-cerebral hemorrhage stroke. We will also exclude patients who have been incapacitated to an extent that they are unable to comprehend a conversation or communicate effectively in a group setting. Additionally, patients will be excluded if they are discharged to a nursing home or who will move out of the New York City area after discharge.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2002-09; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Identification of under-use of effective secondary stroke preventive measures.

SECONDARY OUTCOMES:
Identification of the causes of under-use of effective secondary stroke preventive measures
the characteristics of those patients

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chassin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States